CLINICAL TRIAL: NCT03062241
Title: Cryoablation of Atrial Fibrillation in Patients With Severe Heart Failure
Brief Title: Ablation of Atrial Fibrillation in Heart Failure Patients
Acronym: CONTRA-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Collaborators: Military Institute od Medicine National Research Institute (Other); Clinical Hospital No. 2 Pomeranian Medical University, Szczecin, Poland (Unknown); Hospital name Pope John Paul, Zamosc, Poland (Unknown)
Responsible Party: Principal Investigator, Zbigniew Kalarus, Head of Cardiology Department, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONTRA-HF study
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation; Severe Heart Failure
Keywords: cryoablation; conventional treatment of heart failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: This is a Randomized Controlled Trial (RCT), non-blinded, prospective, multicentre performed in up to 4 cardiology centers in Poland. All patients implanted with a dual-chamber implanted cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D) with Home Monitoring capabilities and history of paroxysmal, persistent or persistant long-lasting AF will be screened for the study. In patient who fulfill all inclusion and none of the exclusion criteria 1 year after ICD or CRT-D implantation, with exclusion of 1 month directly after implantation, a device check-up and AF burden will be performer and assessed. Randomization will be performed using sealed envelopes and will be conducted in the coordinating center of the study PI in all patients who sign informed consent and met all inclusions and none of the exclusion criteria. The cryoablation of AF will be performed within 1 month from randomization in the invasive treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation (Experimental): The pulmonary vein (PV) isolation in patients randomized to intervention group.
  Interventions: Procedure: Cryoablation
- Conventional treatment (No Intervention): Pharmacological treatment according to 2016 ESC (European Society of Cardiology) guidelines for the diagnosis and treatment of acute and chronic heart failure and to 2016 ESC guidelines for the management of atrial fibrillation developed in collaboration with European Association for Cardio-Thoracic Surgery (EACTS).

INTERVENTIONS:
Procedure: Cryoablation — After left atrial appendage (LAA) thrombus exclusion, the transseptal puncture will be performed and intravenous heparin will be administered to achieve Activated Clotting Time (ACT) ≥300 seconds.The pulmonary vein (PV) isolation will be performed. Optimal cryoballoon positioning will be confirmed by PVs angiography. Pulmonary veins isolation will be confirmed by entrance/exit block using appropriate catheter. During cryoablation of the right PVs, high-output right phrenic nerve stimulation will be performed using a diagnostic catheter placed in the superior vena cava. Whenever decrease/loss of pacing capture will be observed, cryoablation will be immediately terminated.
  Arms: Cryoablation

SUMMARY:
The aim of the study is to evaluate the impact of cryoablation of atrial fibrillation in patients with severe chronic heart failure (CHF) on long term outcome of CHF and efficacy (endurance) of the procedure itself. The study hypothesis is that cryoablation in eligible patients with CHF and ICD/CRT (implantable cardioverter defibrillator / cardiac resynchronization therapy) implants reduce the number of recurrent CHF hospitalizations, mortality, need for mechanical support of LV (left ventricle) and heart transplant (primary endpoint) at 1 year observation in comparison to traditional (pharmacological) treatment..

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common arrhythmia worldwide and the risk of AF incidence increases with age. The amount of patients suffered from AF is still underestimated due to insufficient diagnosing silent AF. The incidence of patients with silent, asymptomatic AF might be approx. 80% , particularly in patients with heart failure. The most frequent consequence of undiagnosed AF is not only thromboembolism but also heart failure development and loss of quality of life. The incidence of chronic heart failure (CHF), which is the most frequent consequence of coronary heart disease, still increases and nowadays in patients above 70 years affects approx.10%. What is more, AF which is one of the result of CHF occurred in 30% of those patients. Atrial fibrillation ablation is one of the most established method to treat symptomatic patients and its' efficacy is about 70 - 90 %. Hence, the appropriate and effective treatment of those patients might influence not only on the survival but also the quality of life and functionality of health care system.

Among many data about AF in patients with impaired LV (left ventricle) systolic function there is still a lack of randomized, multicenter trials which would compare the influence of AF cryoablation with conventional treatment in patients with LVEF (left ventricle ejection fraction) ≤ 35% (despite optimal pharmacotherapy) on long term survival and efficacy. The deficiency in this field was an inspiration to conduct this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age ≤ 75 years
* optimal pharmacotherapy within the last 3 months
* New York Heart Association (NYHA) II- IV (out-patient) within the last 3 months
* AF paroxysmal, persistent or persistant long-lasting
* at least 1 episode of paroxysmal AF with the duration of ≥ 30 s or AF burden ≥ 10% during 1 month up to 1 year since ICD or CRT-D implantation
* signed informed consent

Exclusion Criteria:

* age < 18 years or > 75 years
* permanent AF
* contraindications to oral anticoagulation or heparin
* prior AF ablation
* chronic kidney disease requiring dialysis
* untreated hypo- or hyperthyroidism
* breast feeding
* pregnancy
* decompensated heart failure within the last 90 days requiring pressor infusion
* stroke within the last 3 months
* myocardial infarction within the last 3 months
* PCI or CABG within the last 3 months
* active myocarditis
* artificial valve replacement surgery
* severe mitral or aortic stenosis
* coronary artery disease requiring revascularization
* heart transplant
* participation in another study
* comorbidities with expected survival less than 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of hospitalization due to heart failure worsening, mortality, use of mechanical left ventricle support and heart transplant. | one year
  percentage of patients who required intravenous diuretic or pressor administration
Composite outcome of hospitalization due to heart failure worsening, mortality, use of mechanical left ventricle support and heart transplant. | one year
  percentage of patients who died
Composite outcome of hospitalization due to heart failure worsening, mortality, use of mechanical left ventricle support and heart transplant. | one year
  percentage of patients who required mechanical left ventricle support
Composite outcome of hospitalization due to heart failure worsening, mortality, use of mechanical left ventricle support and heart transplant. | one year
  percentage of patients who had a heart transplant

SECONDARY OUTCOMES:
Percentage of patients who had ischaemic cerebral stroke during 12 months follow up | one year
  ischaemic cerebral stroke confirmed in computed tomography

OTHER OUTCOMES:
Percentage of patients with arrhythmias incidence | one year
  the effectiveness of the cryoablation assessed on the device interrogation; atrial fibrillation burden at least 30 seconds
Percentage of patients with arrhythmias incidence | one year
  the effectiveness of the cryoablation assessed on the clinical symptoms; the presence of arrhythmias' related symptoms
Quality of life assessment | one year
  The Minnesota Living with Heart Failure Questionnaire
Left ventricle ejection fraction assessment | one year
  transthoracic echocardiography
Patient capacity assessment | six months
  six minute walk test
Oxygen consumption assessment | six months
  cardio-pulmonary exercise test
Percentage of patients requiring hospitalization because of arrhythmias' incidence or symptoms (atrial fibrillation/ atrial flutter) | one year
  patients who required pharmacological or electrical cardioversion
Percentage of biventricular pacing assessment | one year
  the percentage of biventricular pacing assessed on the device interrogation

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Kalarus, MD, Ph.D., Principal Investigator — Department of Cardiology, Congenital Heart Diseases and Electrotherapy Medical University of Silesia, Silesian Center of Heart Diseases
Locations (1):
- Department of Cardiology, Congenital Heart Diseases and Electrotherapy Medical University of Silesia, Silesian Center of Heart Diseases, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xiong Q, Proietti M, Senoo K, Lip GY. Asymptomatic versus symptomatic atrial fibrillation: A systematic review of age/gender differences and cardiovascular outcomes. Int J Cardiol. 2015 Jul 15;191:172-7. doi: 10.1016/j.ijcard.2015.05.011. Epub 2015 May 7. PMID 25974193
- [Background] Vaidya K, Arnott C, Russell A, Masson P, Sy RW, Patel S. Pulmonary Vein Isolation Compared to Rate Control in Patients with Atrial Fibrillation: A Systematic Review and Meta-analysis. Heart Lung Circ. 2015 Aug;24(8):744-52. doi: 10.1016/j.hlc.2015.02.025. Epub 2015 Mar 14. PMID 25890871
- [Background] Lenarczyk R, Jedrzejczyk-Patej E, Szulik M, Mazurek M, Podolecki T, Kowalczyk J, Kowalski O, Sredniawa B, Kalarus Z; Triple-Site Versus Standard Cardiac Resynchronization Trial (TRUST CRT) Investigators. Atrial fibrillation in cardiac resynchronization recipients with and without prior arrhythmic history. How much of arrhythmia is too much? Cardiol J. 2015;22(3):267-75. doi: 10.5603/CJ.a2014.0102. Epub 2015 Jan 7. PMID 25563708
- [Background] Marrouche NF, Brachmann J; CASTLE-AF Steering Committee. Catheter ablation versus standard conventional treatment in patients with left ventricular dysfunction and atrial fibrillation (CASTLE-AF) - study design. Pacing Clin Electrophysiol. 2009 Aug;32(8):987-94. doi: 10.1111/j.1540-8159.2009.02428.x. PMID 19659616
- [Result] Khan MN, Jais P, Cummings J, Di Biase L, Sanders P, Martin DO, Kautzner J, Hao S, Themistoclakis S, Fanelli R, Potenza D, Massaro R, Wazni O, Schweikert R, Saliba W, Wang P, Al-Ahmad A, Beheiry S, Santarelli P, Starling RC, Dello Russo A, Pelargonio G, Brachmann J, Schibgilla V, Bonso A, Casella M, Raviele A, Haissaguerre M, Natale A; PABA-CHF Investigators. Pulmonary-vein isolation for atrial fibrillation in patients with heart failure. N Engl J Med. 2008 Oct 23;359(17):1778-85. doi: 10.1056/NEJMoa0708234. PMID 18946063
- [Result] Zhao L, Xu K, Jiang W, Zhou L, Wang Y, Zhang X, Wu S, Liu X. Long-term outcomes of catheter ablation of atrial fibrillation in dilated cardiomyopathy. Int J Cardiol. 2015;190:227-32. doi: 10.1016/j.ijcard.2015.04.186. Epub 2015 Apr 23. PMID 25920033
- [Result] Bunch TJ, May HT, Bair TL, Jacobs V, Crandall BG, Cutler M, Weiss JP, Mallender C, Osborn JS, Anderson JL, Day JD. Five-year outcomes of catheter ablation in patients with atrial fibrillation and left ventricular systolic dysfunction. J Cardiovasc Electrophysiol. 2015 Apr;26(4):363-370. doi: 10.1111/jce.12602. Epub 2015 Feb 11. PMID 25534572
- [Result] Rillig A, Makimoto H, Wegner J, Lin T, Heeger C, Lemes C, Fink T, Metzner A, Wissner E, Mathew S, Wohlmuth P, Kuck KH, Tilz RR, Ouyang F. Six-Year Clinical Outcomes After Catheter Ablation of Atrial Fibrillation in Patients With Impaired Left Ventricular Function. J Cardiovasc Electrophysiol. 2015 Nov;26(11):1169-1179. doi: 10.1111/jce.12765. Epub 2015 Sep 3. PMID 26217925
- [Result] Schwartzman D, Housel D, Bazaz R, Jain S, Saba S, Gorcsan J 3rd, Adelstein E. A pilot study to assess benefit of atrial rhythm control after cardiac resynchronization therapy and atrioventricular node ablation. Pacing Clin Electrophysiol. 2015 Feb;38(2):275-81. doi: 10.1111/pace.12535. Epub 2014 Nov 27. PMID 25431023